CLINICAL TRIAL: NCT05570500
Title: Comparing the Effect of the Online Oral Health Education to the Conventional Method on the Knowledge and Practice of Personal Oral Hygiene in a Group of Primary School Children in Egypt. A Randomized Controlled Trial
Brief Title: Comparing the Effect of Online and Conventional Oral Health Education in Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar Alaa Taqa, Master's degree student, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DPH20-3M
Record Dates: First submitted 2022-09-22; First posted 2022-10-06 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Knowledge; Attitude to Health; Practice
Keywords: oral health education; oral health promotion; school children
MeSH Terms: interventions — Health Education, Dental

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the participants will know the group they are assigned to since they need to access the online oral health education sessions in case of being assigned to that group. The participants in conventional method will receive their oral health education sessions in their classrooms directly, thus making it impossible to mask both participant groups.
  the care provider is the primary investigator, and he is the person responsible of delivering the oral health education sessions which makes it impossible to mask the intervention details.
  Only the outcomes assessor (which is the statistician) will be blinded from the groups involved, names of participants and study details.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group, conventional oral health education group (Placebo Comparator)
  Interventions: Behavioral: Oral health education
- Comparison group, online oral health education group (Active Comparator)
  Interventions: Behavioral: Oral health education

INTERVENTIONS:
Behavioral: Oral health education — oral health education sessions that aims to improve both knowledge of primary school children regarding bacteria, caries, number of teeth, plaque formation and attitude of primary school children regarding tooth brushing techniques, number of times per day, dietary instructions to avoid dental caries.

SUMMARY:
This study aims to compare the results of online oral health education and conventional oral health education methods in terms of their effectiveness towards improving the knowledge and practice of oral hygiene in primary school children in Egypt.

This study is done in two schools in Egypt, in 3rd and 4th grade respectfully. The classrooms in each grade will be randomly assigned to each of the two groups (online and conventional oral health education). A questionnaire that assesses knowledge and attitude towards self oral care will be administered by the primary investigator before and after the oral health education sessions. The pre and post questionnaires will be compared in terms of results to evaluate the effectiveness of both methods.

ELIGIBILITY:
Inclusion Criteria:

* 3rd and 4th grade Egyptian students.
* Average of age 7-10 years old.
* Currently residing in Egypt.
* Both male and female students.

Exclusion Criteria:

* Those who do not consent to participate in the study.
* Those who cannot speak English or Arabic.
* Non-Egyptians

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 636 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amira S Badran, PHD, Study Director — Ain Shams University; Omar A Taqa, student, Principal Investigator — Ain Shams University
Locations (1):
- Futures language schools, Cairo, Sherook Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO, EMRO (2014, September 3). WHO EMRO | Egypt releases results of epidemiological study on oral health status. Available from: http://www.emro.who.int/egy/egypt-events/results-of-epidemiological-study-on-oral-health-status-released.html
- [Background] Mohamed, yomna. (2020). Assessment of the Knowledge and Awareness Among Egyptian Parents in Relation To Oral Health Status of Their Children. Egyptian Dental Journal, 66(2), 737-746. https://doi.org/10.21608/edj.2020.25196.1058
- [Background] Gambhir RS, Sohi RK, Nanda T, Sawhney GS, Setia S. Impact of school based oral health education programmes in India: a systematic review. J Clin Diagn Res. 2013 Dec;7(12):3107-10. doi: 10.7860/JCDR/2013/6212.3718. Epub 2013 Dec 15. PMID 24551745
- [Background] Alsumait A, ElSalhy M, Amin M. Long-Term Effects of School-Based Oral Health Program on Oral Health Knowledge and Practices and Oral Health-Related Quality of Life. Med Princ Pract. 2015;24(4):362-8. doi: 10.1159/000430096. Epub 2015 Jun 2. PMID 26045154
- [Background] 5- WHO (2020) Timeline: WHO's COVID-19 response. Available from: https://www.who.int/emergencies/diseases/novel-coronavirus-2019/interactive-timeline?gclid=Cj0KCQjwufn8BRCwARIsAKzP6964UmFJZqWX9mc0tE7Fu5DVDnlzOskefX9AJAtBy8zOdgnZqtCPK3gaAoUhEALw_wcB
- [Background] 6- WHO (2020) health topics / coronavirus. Available from: https://www.who.int/health-topics/coronavirus#tab=tab_1
- [Background] 7- Ayoub, G. M. (2019). Teachers' experiences in overcrowded classrooms in Egyptian public schools.
- [Background] 8- Egyptian ministry of education online portal. Available from: http://portal.moe.gov.eg/eng/Pages/default.aspx#
- [Background] Kwan SY, Petersen PE, Pine CM, Borutta A. Health-promoting schools: an opportunity for oral health promotion. Bull World Health Organ. 2005 Sep;83(9):677-85. Epub 2005 Sep 30. PMID 16211159
- [Background] Angelopoulou MV, Kavvadia K, Taoufik K, Oulis CJ. Comparative clinical study testing the effectiveness of school based oral health education using experiential learning or traditional lecturing in 10 year-old children. BMC Oral Health. 2015 Apr 28;15:51. doi: 10.1186/s12903-015-0036-4. PMID 25924670
- [Background] GeethaPriya PR, Asokan S, Kandaswamy D, Shyam S. Impact of different modes of school dental health education on oral health-related knowledge, attitude and practice behaviour: an interventional study. Eur Arch Paediatr Dent. 2020 Jun;21(3):347-354. doi: 10.1007/s40368-019-00489-7. Epub 2019 Nov 16. PMID 31734931
- [Background] Cascaes AM, Bielemann RM, Clark VL, Barros AJ. Effectiveness of motivational interviewing at improving oral health: a systematic review. Rev Saude Publica. 2014 Feb;48(1):142-53. doi: 10.1590/s0034-8910.2014048004616. PMID 24789647
- [Background] 13- Miller, W. R., & Rollnick, S. (2002). Motivational interviewing: Preparing people for change (2nd ed.). The Guilford Press.
- [Background] Gao X, Lo EC, McGrath C, Ho SM. Face-to-face individual counseling and online group motivational interviewing in improving oral health: study protocol for a randomized controlled trial. Trials. 2015 Sep 18;16:416. doi: 10.1186/s13063-015-0946-0. PMID 26385340
- [Background] 15- Acharya, Sonu. (2019). Motivational Interviewing in Pediatric Dentistry: Role in Behavior Management. Journal of South Asian Association of Pediatric Dentistry. 2. 69-72. 10.5005/jp-journals-10077-3030.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Classrooms
Groups:
- Comparison Group, Online Oral Health Education Group: In this study group, participants received online oral health education session by logging in their Microsoft teams accounts.
  The intervention applied during the online oral health education session was in a form of pre-recorded cartoon presentation created by Prezi software.
- Control Group, Conventional Oral Health Education Group: In this study group, participants received face-to-face oral health education session live inside their classrooms.
  The intervention applied during the conventional oral health education session was a live demo on toothbrushing techniques and a cartoon presentation created by using Prezi software.
Period: Overall Study
Arm/Group | Comparison Group, Online Oral Health Education Group | Control Group, Conventional Oral Health Education Group
Started | 319; 8 Classrooms (This is the total number of participants (children) in the online oral health education group, divided into 150 males and 169 females in this study group.) | 317; 8 Classrooms (This is the total number of participants (children) in the conventional oral health education group, divided into 155 males and 162 females in this study group.)
Classroom 1 in Each Study Group | 42; 1 Classrooms | 40; 1 Classrooms
Classroom 2 in Each Study Group | 38; 1 Classrooms | 39; 1 Classrooms
Classroom 3 in Each Study Group | 39; 1 Classrooms | 41; 1 Classrooms
Classroom 4 in Each Study Group | 36; 1 Classrooms | 42; 1 Classrooms
Classroom 5 in Each Study Group | 41; 1 Classrooms | 37; 1 Classrooms
Classroom 6 in Each Study Group | 40; 1 Classrooms | 39; 1 Classrooms
Classroom 7 in Each Study Group | 43; 1 Classrooms | 41; 1 Classrooms
Classroom 8 in Each Study Group | 40; 1 Classrooms | 38; 1 Classrooms
Completed | 312; 8 Classrooms | 312; 8 Classrooms
Not Completed | 7; 0 Classrooms | 5; 0 Classrooms
Not completed — Lost to Follow-up | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group, Conventional Oral Health Education Group | Comparison Group, Online Oral Health Education Group | Total
Number analyzed (Participants) | 312 | 312 | 624
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 312 | 312 | 624
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 150 | 315
  Male | 147 | 162 | 309
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 312 | 312 | 624

OUTCOME MEASURES:

1. Primary Outcome: Effect of Oral Health Education on the Oral Health Knowledge in Primary School Children Aged 7-9 Years Old
Description: A questionnaire will be assigned to the participants to determine level of knowledge. Higher mean value of correct answer is considered to be of satisfactory outcome. lesser mean value of correct answers is considered to be unsatisfactory.
  The scale of measurement would be the total number of scores per participant entry on the knowledge section of the questionnaire. The knowledge section of the questionnaire contains 5 questions, 4 single answer questions and 1 multiple-answer question with two correct answers. The total score for the knowledge section is 6 marks (4+2), where the lowest score is 0 and the highest is 6. Higher scores mean better outcomes and lower scores mean worse outcomes.
Time Frame: 2 months
Population: all participants in both arms received oral health education session through colorful images and cartoons.
Measure: Mean (Standard Deviation); unit: knowledge score on a scale
Arm/Group | Control Group, Conventional Oral Health Education Group | Comparison Group, Online Oral Health Education Group
Number analyzed (Participants) | 312 | 312
knowledge score on a scale | 2.71 (1.53) | 0.81 (1.16)

2. Secondary Outcome: Effect of Oral Health Education on Oral Hygiene Measures Practice in Primary School Children Aged 7-9 Years Old
Description: A questionnaire will be assigned to the participants to determine the practice level of children towards oral hygiene. The scale of measurement would be on a percentage of correct answers, with minimum value denoting 0% and maximum value of 100%. Higher scores mean better outcomes and lower scores mean worse outcomes.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group, Conventional Oral Health Education Group | Comparison Group, Online Oral Health Education Group
Number analyzed (Participants) | 312 | 312
Participants
  participants who brushed their teeth two times or more | 224 | 208
  participants who brushed less than two times or forgot to brush their teeth | 84 | 97
  participants who dont brush their teeth | 4 | 7

ADVERSE EVENTS:
Description: Death, serious adverse events and other (non-serious adverse events) were not assessed for the study
Groups:
- Control Group, Conventional Oral Health Education Group: Participants in this group received oral health education in their classrooms. The oral health education session included a demo on toothbrushing techniques and a cartoon presentation showing dental caries process.
  Oral health education sessions are sessions that aim to improve both knowledge of primary school children regarding bacteria, caries, number of teeth, plaque formation and attitude of primary school children regarding tooth brushing techniques, number of times per day, dietary instructions to avoid dental caries.
- Comparison Group, Online Oral Health Education Group: Participants in this group received oral health education sessions by logging in their Microsoft teams accounts and accessing the presentation which was created using Prezi software. The presentation included visual cartoons on dental caries process and toothbrushing techniques.
  Oral health education sessions are sessions that aim to improve both knowledge of primary school children regarding bacteria, caries, number of teeth, plaque formation and attitude of primary school children regarding tooth brushing techniques, number of times per day, dietary instructions to avoid dental caries.
Arm/Group | Control Group, Conventional Oral Health Education Group | Comparison Group, Online Oral Health Education Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-11-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05570500/Prot_000.pdf